CLINICAL TRIAL: NCT03146897
Title: Comparison of Four Different Supplementary Foods in the Treatment of Moderate Acute Malnutrition (MAM) in Children: Sierra Leone Cost-Effectiveness Study
Brief Title: Comparison of Four Different Supplementary Foods in the Treatment of Moderate Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Washington University School of Medicine (Other); Project Peanut Butter (Other); Caritas Bo (Unknown); Ministry of Health and Sanitation, Sierra Leone (Other Government); United Nations World Food Programme (WFP) (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lindsey Green, Beatrice Lorge Rogers, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAQR
Record Dates: First submitted 2017-04-13; First posted 2017-05-10 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Moderate Acute Malnutrition
Keywords: Food Aid, Malnutrition, RUSF, FBF, Supplementary Food
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Super Cereal Plus with amylase (Active Comparator)
  Interventions: Dietary Supplement: Supplementary Food
- Corn-soy Blend Plus and Vegetable Oil (Active Comparator)
  Interventions: Dietary Supplement: Supplementary Food
- Corn-soy Whey Blend and Vegetable Oil (Active Comparator)
  Interventions: Dietary Supplement: Supplementary Food
- Ready-to-Use-Supplementary Food (Active Comparator)
  Interventions: Dietary Supplement: Supplementary Food

INTERVENTIONS:
Dietary Supplement: Supplementary Food — Supplementary food for treating MAM

SUMMARY:
The research seeks to determine the relative effectiveness and cost effectiveness of alternative supplementary foods in the treatment of moderate acute malnutrition (MAM) in normal program settings. The results of this study will guide decisions about what commodities to use in supplementary feeding programs in particular contexts and populations, and what factors need to be addressed to ensure maximum effectiveness in the treatment of moderate malnutrition.

Tufts University, Washington University in St. Louis, School of Medicine, Sierra Leone Ministry of Health and Sanitation (MoHS), Project Peanut Butter, Caritas Bo, World Food Programme (WFP), and the United States Agency for International Development (USAID) are collaborating to conduct an assessment of the effectiveness, cost, and cost-effectiveness of food aid commodities in treating moderate acute malnutrition (MAM) in young children. The study comparison is based on a targeted food delivery to children 6-59 months who are screened for MAM. Study participants will receive one of four approximately isoenergetic test foods:

1. Super Cereal Plus (SC+) with amylase
2. Corn-soy Blend Plus (CSB+) and fortified vegetable oil
3. Corn-soy Whey Blend (CSWB) and fortified vegetable oil (CSWB is a new product which is a modified version of CSB)
4. Ready-to-use Supplementary Food (RUSF, lipid-based)

DETAILED DESCRIPTION:
The proposed research seeks to determine the relative effectiveness and cost effectiveness of alternative supplementary foods in the treatment of moderate acute malnutrition (MAM) in normal program settings. The results of this study will guide decisions about what commodities to use in supplementary feeding programs in particular contexts and populations, and what factors need to be addressed to ensure maximum effectiveness in the treatment of moderate malnutrition.

Tufts University, Washington University in St. Louis, School of Medicine, Sierra Leone Ministry of Health and Sanitation (MoHS), Project Peanut Butter, Caritas Bo, World Food Programme (WFP), and the United States Agency for International Development (USAID) are collaborating to conduct an assessment of the effectiveness, cost, and cost-effectiveness of food aid commodities in treating moderate acute malnutrition (MAM) in young children. The study comparison is based on a targeted food delivery to children 6-59 months who are screened for MAM. Study participants will receive one of four approximately isoenergetic test foods:

1. Super Cereal Plus (SC+) with amylase
2. Corn-soy Blend Plus (CSB+) and fortified vegetable oil
3. Corn-soy Whey Blend (CSWB) and fortified vegetable oil (CSWB is a new product which is a modified version of CSB)
4. Ready-to-use Supplementary Food (RUSF, lipid-based)

Type of study: This will be a prospective, cluster-randomized, controlled clinical effectiveness trial.

Peripheral Health Units (PHU) will be selected within the Pujehun District in Sierra Leone. These 29 PHUs and the villages they serve will be used as the study sites to test the effectiveness of four supplementary foods in the treatment of MAM. The PHUs will be grouped into 4 to represent each food or arm of the study. The study is targeting 6000 children in total: 1500 children per arm. Children will be enrolled and graduated based on mid-upper arm circumference (MUAC); weight and height will be recorded as well and also used in final analysis. Locations (communities, clinics) will be assigned to one of the four arms (that is, foods to be tested). The foods distributed as part of the study will require a safe storage location.

Supplementary food rations will be delivered for up to 12 weeks from enrollment (enrollment takes place when a child is diagnosed with MAM in accordance with a mid-upper-arm-circumference [MUAC] >11.5 cm and ≤12.5 cm). Children will be asked to return to the PHU every two weeks for follow-up, where caretakers report on the child's clinical symptoms and use of the food at home, growth measurements are re-assessed, until they reach one of the primary outcomes listed below. A ration of supplementary food sufficient for two weeks (14 days) will be distributed at each visit. Children will be monitored for relapse after discharge and be interviewed for basic IYCF information at graduation, 1-month and 3-month follow up.

The primary outcome measures are graduation from MAM (achieving MUAC ≥ 12.5 cm by 12 weeks) once or failure (death, development of severe acute malnutrition, transfer to hospital for inpatient care, failure to graduate from MAM by 12 weeks, default).

Additional analysis will consider achievement of WHZ => -2 among children treated for either up to 12 weeks or until reaching graduation based on MUAC. Secondary outcome measures include rates of weight, height, and MUAC gain, change in WHZ, LAZ, and HAZ , WHZ ≥ -2, time to graduation, and any possible adverse effects from the supplementary foods.

Cost effectiveness will assess differences among the four study arms in cost per case of MAM graduated.

The field research team will randomly select a subsample of caregivers of enrolled children for in-depth interviews and in-home observations, which will take place in the participants' home. In addition, the field research team will conduct focus group discussions with a smaller subsample of caregivers, to take place in a central and convenient location. The purpose of the in-home observations is to observe aspects of the family's preparation and consumption of the ration that they would be unlikely to be able to report during focus groups or individual interviews, because respondents may not be conscious of their actions. We will also collect data on behaviors, demographics and other factors contributing to effectiveness, including: ration collection, preparation, consumption, sharing, and selling behaviors, knowledge and communication of social and behavior change communication (SBCC) messages regarding ration use among health workers and beneficiary mothers, other health behaviors such as breastfeeding, dietary diversity and hygiene practices, and demographics such as household food insecurity and number of young children. All interviews, observations, and focus group discussions will be administered by trained research assistants. The team will also conduct interviews with community health volunteers working in the PHUs and the catchment villages they serve.

The research team will implement three sub-studies that aim to:

1. Compare the effect of four supplementary foods on changes in body composition of 6-59 month-old children with MAM after four weeks of treatment.
2. Examine whether EED modifies the effect of four supplementary foods on 6-59 month-old children with MAM.
3. Examine the effects of MAM and 4 supplementary foods on neurocognitive function in 6-24 month-old children.

This study will benefit the food assistance community by providing new research on the cost and cost-effectiveness of supplements to treat MAM, where effectiveness is measured in terms of growth outcomes.

Besides the long term and broader benefits, this work will benefit a large number of young children in the Sierra Leone population. This study will directly benefit Sierra Leone by improving the nutrition of its children and providing education on children's nutrition. The enrolled child will have enough study food provided at home for the recovery from moderate acute malnutrition when consumed along with the regular diet and will be monitored regularly during treatment. This may result in fewer complications (diarrhea, respiratory illnesses) as the child recovers.

ELIGIBILITY:
Inclusion Criteria:

* Child diagnosed with MAM based on MUAC and enrolled to receive a ration from a feeding site (i.e. enrolled in the SFP)

Exclusion Criteria:

* Children with bipedal oedema
* Children receiving food rations from another organization (e.g. USAID, WFP, UNICEF) for treatment of MAM
* Children who have previously been enrolled in the study (they are not eligible to be re-enrolled in the study but are still eligible to receive food)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2691 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-11-24 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness assessed by recovery from MAM, defined as achieving mid-upper arm circumference (MUAC) ≥ 12.5 cm within the 12-week treatment period | 12 weeks
  Graduation from MAM, defined as achieving mid-upper arm circumference (MUAC) ≥ 12.5 cm within the 12-week treatment period
Cost-Effectiveness | 12 weeks
  Assess program costs among the four study arms including fixed, start-up and ongoing costs of food supplements, repackaging, transportation, storage, distribution, other clinical and SBCC programming activities, and caregivers' opportunity costs. Link these costs with the effectiveness outcomes to determine and compare the cost-effectiveness of using each supplement to treat MAM (e.g. Cost per Case of MAM graduated).
WHZ => -2 SD among children treated for up to 12 weeks or until reaching graduation based on MUAC whose WHZ was < -2 SD at enrollment | 12 weeks
  Percent of children enrolled in MAM treatment whose WHZ => -2 SD (calculated based on height at enrollment and weight at graduation) at graduation based on MUAC or at 12 weeks of treatment, whichever is earliest, taking into consideration their WHZ at enrollment.

SECONDARY OUTCOMES:
Weight (g/kg/d) | 4 weeks
  Weight (g/kg/d)
MUAC (mm/d) gain within first 4 weeks | 4 weeks
  MUAC (mm/d) gain within first 4 weeks
Change in weight-for-height Z score (WHZ) and height-for-age Z score (HAZ), height gain (mm/d), enrollment to discharge and 1,3,6 months post discharge | 6 months
  Change in weight-for-height Z score (WHZ) and height-for-age Z score (HAZ), height gain (mm/d), enrollment to discharge and 1,3,6 months post discharge
Time to graduation | 12 weeks
  Time to graduation (for those who graduated)
Post-treatment growth status | Up to 6 months after graduation/discharge
  Post-treatment growth status at 1, 3, and 6 months after graduation/discharge.
Achieving WHZ >= -2 SD (using weight at the last visit and length at admission) at discharge and at 1,3 and 6 months post discharge | Up to 6 months after graduation/discharge
  Achieving WHZ >= -2 SD (using weight at the last visit and length at admission) at discharge and at 1,3 and 6 months post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Rogers, PhD, Principal Investigator — Tufts University; Mark Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Stacy Griswold, MS, Pujehun, Sierra Leone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griswold SP, Langlois BK, Shen Y, Cliffer IR, Suri DJ, Walton S, Chui K, Rosenberg IH, Koroma AS, Wegner D, Hassan A, Manary MJ, Vosti SA, Webb P, Rogers BL. Effectiveness and cost-effectiveness of 4 supplementary foods for treating moderate acute malnutrition: results from a cluster-randomized intervention trial in Sierra Leone. Am J Clin Nutr. 2021 Sep 1;114(3):973-985. doi: 10.1093/ajcn/nqab140. PMID 34020452
- [Derived] Suri DJ, Potani I, Singh A, Griswold S, Wong WW, Langlois B, Shen Y, Chui KHK, Rosenberg IH, Webb P, Rogers BL. Body Composition Changes in Children during Treatment for Moderate Acute Malnutrition: Findings from a 4-Arm Cluster-Randomized Trial in Sierra Leone. J Nutr. 2021 Jul 1;151(7):2043-2050. doi: 10.1093/jn/nxab080. PMID 33880554